CLINICAL TRIAL: NCT01516255
Title: A Thorough QTc Evaluation of the Effect of Liraglutide on Cardiac Repolarization in Healthy Volunteers: A Randomized, Double-blind, Placebo-controlled, Two Period Crossover Study Followed by Open-label Moxifloxacin (Positive Control) Administration
Brief Title: Effect of Liraglutide on Heart Frequency in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1644
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Double-blind / liraglutide (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo; Procedure: electrocardiogram (ECG)
- Double-blind / placebo (Placebo Comparator)
  Interventions: Drug: liraglutide; Drug: placebo; Procedure: electrocardiogram (ECG)
- Open-label / moxifloxacin (Active Comparator)
  Interventions: Drug: moxifloxacin; Procedure: electrocardiogram (ECG)
- Open-label / placebo (Placebo Comparator)
  Interventions: Drug: placebo; Procedure: electrocardiogram (ECG)

INTERVENTIONS:
Drug: liraglutide — 0.6 mg daily for 7 days followed by 1.2 mg daily for 7 days followed by 1.8 mg daily for 7 days. Injected subcutaneously. Subjects are randomly allocated to two treatment sequences
  Arms: Double-blind / liraglutide; Double-blind / placebo
Drug: placebo — Injected subcutaneously. Subjects are randomly allocated to two treatment sequences
  Arms: Double-blind / liraglutide; Double-blind / placebo
Drug: moxifloxacin — Following the double-blinded period and a wash-out period of 7 days, subjects are re-randomised to an open-label, parallel period where a single dose of 400 mg moxifloxacin (tablets) is administered as positive control
  Arms: Open-label / moxifloxacin
Drug: placebo — Following the double-blinded period and a wash-out period of 7 days, subjects are re-randomised to an open-label, parallel period where single dose of oral placebo is administered
  Arms: Open-label / placebo
Procedure: electrocardiogram (ECG) — 24 hours serial ECG is collected before initial dose of 0.6 mg liraglutide, on the last dosing day of 1.2 mg liraglutide and on the last dosing day of 1.8 mg liraglutide
  Arms: Double-blind / liraglutide; Double-blind / placebo
Procedure: electrocardiogram (ECG) — Six hours after moxifloxacin or placebo single dose, 1 hour serial ECG is collected
  Arms: Open-label / moxifloxacin; Open-label / placebo

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to investigate if liraglutide effects the QTc interval. Moxifloxacin (Avelox®) is administered as positive control.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Fasting plasma glucose within normal limits (80-100 mg/dl)
* BMI (Body Mass Index): 20.0-29.0 kg/m^2 (inclusive)
* Heart rate within the range of 50-90 beats per minute (inclusive)
* Subject is judged to be in good health on the basis of their medical history, physical examination, ECG (electrocardiogram), and routine laboratory data

Exclusion Criteria:

* Any clinically significant disease history, in the opinion of the investigator, of systemic or organ disease
* Any clinically significant disease history, in the opinion of the investigator, of cardiovascular disease
* Clinically significant abnormalities on any pre-study clinical examination or any abnormal laboratory measurements during screening
* A family history of sudden cardiac death at age less than 50 years old
* T-wave abnormalities
* Individual or familial history of long QT Syndrome
* Positive results on Screening for Hepatitis B surface antigen, Hepatitis C antibody or HIV (human immunodeficiency virus) antibody
* Positive results on the urine drug and alcohol screen
* Any regular use of prescription or nonprescription drugs or vitamins and herbal/nutritional supplements that cannot be stopped at screening
* Any strenuous exercise (as judged by the investigator) from 4 days prior to randomisation and during the entire trial period
* Blood donation, trauma or surgery with blood loss exceeding 500 ml within the last 2 months prior to dosing
* Subject is a smoker, occasional smoker or has a history of smoking (or use of any tobacco) within the last 3 months
* Excessive use of methylxanthine-containing beverages (more than 8 cups/day of coffee, tea, soda or chocolate)
* Females who are pregnant, breastfeeding, intend to become pregnant within the next 3 months, or who are judged to be using inadequate contraceptive measures
* A history (within the last 2 years) of drug or alcohol abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2006-07; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Maximum time-matched mean difference between the baseline subtracted QTci intervals

SECONDARY OUTCOMES:
QTc at liraglutide tmax (time to reach maximum concentration)
Percentage subjects with QTc at least 450, 480 and 500 milliseconds
Moxifloxacin maximum time-matched mean change QTc and QTci
Cmax, maximum concentration of liraglutide
tmax, time to reach Cmax of liraglutide
Vitals signs: Blood pressure
Vital signs: Pulse
Serial electrocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Fargo, North Dakota, United States

REFERENCES:
- [Result] Chatterjee DJ, Khutoryansky N, Zdravkovic M, Sprenger CR, Litwin JS. Absence of QTc prolongation in a thorough QT study with subcutaneous liraglutide, a once-daily human GLP-1 analog for treatment of type 2 diabetes. J Clin Pharmacol. 2009 Nov;49(11):1353-62. doi: 10.1177/0091270009339189. Epub 2009 Sep 8. PMID 19737980
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com